CLINICAL TRIAL: NCT00023998
Title: A Groupwide Phase II Study of Trastuzumab (Herceptin) in Metastatic Osteosarcoma Patients With Tumors That Overexpress HER2
Brief Title: Chemotherapy With or Without Trastuzumab in Treating Patients With Metastatic Osteosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01863; AOST0121; U10CA098543 (NIH); CDR0000068882 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Metastatic Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Doxorubicin; Cisplatin; Methotrexate; merphos; Leucovorin; Filgrastim; Granulocyte Colony-Stimulating Factor; Radiotherapy; Radiation; Etoposide; Ifosfamide; indolepropanol phosphate; Trastuzumab

ARMS (1):
- Treatment (combination chemotherapy) (Experimental): See detailed description.
  Interventions: Drug: doxorubicin hydrochloride; Drug: cisplatin; Drug: methotrexate; Drug: leucovorin calcium; Biological: filgrastim; Procedure: therapeutic conventional surgery; Radiation: radiation therapy; Drug: etoposide; Drug: ifosfamide; Biological: trastuzumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: methotrexate — Given IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Drug: leucovorin calcium — Given IV or orally
  Other Names: CF; CFR; LV
Biological: filgrastim — Given IV
  Other Names: G-CSF; Neupogen
Procedure: therapeutic conventional surgery — Undergo resection
Radiation: radiation therapy — Undergo radiotherapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Drug: ifosfamide — Given IV
  Other Names: Cyfos; Holoxan; IFF; IFX; IPP
Biological: trastuzumab — Given IV
  Other Names: anti-c-erB-2; Herceptin; MOAB HER2
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as trastuzumab can locate tumor cells and kill them without harming normal cells. Combining monoclonal antibody therapy with chemotherapy may kill more tumor cells. Phase II trial to study the effectiveness of chemotherapy with or without trastuzumab in treating patients who have metastatic osteosarcoma

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the feasibility and safety of trastuzumab (Herceptin) and chemotherapy in patients with HER2-overexpressing (2+ level of expression) metastatic osteosarcoma.

II. Determine the response rate and 3-year event-free survival of patients treated with this regimen.

III. Determine the cardiac toxicity and late effects of this regimen in these patients.

IV. Determine the response rate and 3-year event-free survival of poor-risk patients with HER2-negative tumors treated with chemotherapy without the addition of trastuzumab.

OUTLINE: This is a multicenter study. Patients are stratified according to tumor HER2 status (positive vs negative).

Patients receive induction therapy comprising doxorubicin IV over 20 minutes followed by cisplatin IV over 4 hours on days 1 and 2 of weeks 1 and 6, and methotrexate IV over 4 hours on day 1 of weeks 4, 5, 9, and 10. Patients also receive leucovorin calcium IV or orally every 6 hours beginning 24 hours after each methotrexate dose and continuing for at least 10 doses until methotrexate levels sufficiently decrease. Within 24-36 hours after completion of induction therapy, patients receive filgrastim (G-CSF) daily until blood counts recover.

Patients undergo resection of any remaining primary tumor and/or metastatic lesions during week 11. Patients who are unable to undergo resection receive radiotherapy between weeks 11 and 17.

Patients receive post-induction therapy comprising doxorubicin IV over 20 minutes on days 1 and 2 of weeks 17, 25, and 29; cisplatin IV over 4 hours on days 1 and 2 of weeks 17 and 25; methotrexate IV over 4 hours on day 1 of weeks 16, 20, 24, 28, 32, and 33; etoposide IV over 1 hour on days 1-5 of weeks 13, 21, and 34; and ifosfamide IV over 4 hours on days 1-5 of weeks 13, 21, 29, and 34. Patients also receive leucovorin calcium and G-CSF as in induction therapy. Patients whose tumors are found to over express HER2 (2+ level of expression) also receive trastuzumab IV over 30-90 minutes once a week for a total of 34 weeks in addition to the chemotherapy regimen.

Patients are followed monthly for 1 year, every 2 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 80 patients (40 patients per stratum) will be accrued for this study within 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed high-grade osteosarcoma

  * Metastatic
  * Newly diagnosed
* No osteosarcoma arising in areas of Paget's disease or radiotherapy-induced sarcoma
* Presenting with at least 1 of the following:

  * Bone metastases with or without lung metastases
  * Bilateral lung metastases (any number of nodules)
  * Unilateral lung metastases with at least 4 nodules
* Planned resection of either the primary site or a metastatic site of disease after completion of induction therapy
* Must be currently enrolled on the tumor biology study COG-P9851
* Performance status - ECOG 0-2
* Performance status - Karnofsky 50-100% (over age 10)
* Performance status - Lansky 50-100% (age 10 and under)
* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3
* Bilirubin ≤ 1.5 times normal
* SGPT ≤ 3 times normal
* Creatinine ≤ 1.5 times normal
* Creatinine clearance or glomerular filtration rate ≥ 70 mL/min
* Shortening fraction ≥ 28% by echocardiogram
* Ejection fraction ≥ 50% by echocardiogram or MUGA
* No history of pericarditis, myocarditis, symptomatic arrhythmia, or conduction disturbances
* Normal organ function
* HIV negative
* Not pregnant or nursing
* Fertile patients must use effective contraception
* No prior chemotherapy
* No prior radiotherapy
* See Disease Characteristics

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2001-07; Primary Completion 2005-11 (Actual); Study Completion 2007-05

PRIMARY OUTCOMES:
Feasibility and safety of treatment assessed using CTC version 2.0 | Up to 6 years
  Descriptive statistics will be utilized to assess feasibility and safety. All toxicities will be carefully monitored. A detailed tabulation of observed toxicities will be made and a qualitative decision on the feasibility will be made.
Response rate | Up to 6 years
  Will be estimated with a maximum standard error of no more than 8%.
Event free survival (EFS) | 3 years
  Will be estimated by the Kaplan-Meier method with a maximum standard error of 8%.

CONTACTS AND LOCATIONS:
Overall Officials: David Ebb, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States

REFERENCES:
- [Derived] Kopp LM, Womer RB, Schwartz CL, Ebb DH, Franco VI, Hall D, Barkauskas DA, Krailo MD, Grier HE, Meyers PA, Wexler LH, Marina NM, Janeway KA, Gorlick R, Bernstein ML, Lipshultz SE; Children's Oncology Group. Effects of dexrazoxane on doxorubicin-related cardiotoxicity and second malignant neoplasms in children with osteosarcoma: a report from the Children's Oncology Group. Cardiooncology. 2019 Oct 28;5:15. doi: 10.1186/s40959-019-0050-9. eCollection 2019. PMID 32154021